CLINICAL TRIAL: NCT02707120
Title: Randomized, Parallel Groups, Multicenter and Blind to Evaluators Clinical Trial, to Evaluate the Efficacy and Safety of PRGF-Endoret Eye Drops, in Patients With Stage 2 and 3 Neurotrophic Keratitis
Brief Title: Efficacy and Safety of Plasma Rich in Growth Factors (PRGF-Endoret) Eye-drops in the Treatment of Neurotrophic Keratitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was suspended due to recruitment difficulties
Sponsor: Biotechnology Institute IMASD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTI-011-EC/15/QUER
Record Dates: First submitted 2016-02-29; First posted 2016-03-14 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Neurotrophic Keratitis
Keywords: PRGF, Neurotrophic Keratitis, platelet rich plasma, PRP

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRGF-Endoret eye-drops (Experimental)
  Interventions: Drug: PRGF-Endoret
- Artificial tears eye-drops (Active Comparator)
  Interventions: Drug: Artificial tears eye-drops

INTERVENTIONS:
Drug: PRGF-Endoret — Active treatment will be PRP eye drops obtained by the PRGF-Endoret system.
  Arms: PRGF-Endoret eye-drops
Drug: Artificial tears eye-drops — Artificial tear moisturizing eyedrops (Hidrathea®, Nacl 0.9 % solution without preservatives).
  Arms: Artificial tears eye-drops

SUMMARY:
Neurotrophic keratitis (NK) is a rare degenerative corneal disease caused by altered innervation of the trigeminal nerve that leads to rupture of the corneal epithelium, the regeneration deterioration and development of corneal ulceration, their fusion, and perforation The main characteristic in the NK is a decrease or absence of corneal sensitivity.

DETAILED DESCRIPTION:
The goals of treatment in the neurotrophic keratitis are prevent the progression of corneal damage, maintain eye structure and improve the transparency of the cornea. Therapy should be initiated early and based on the clinical stage of the disease because it depends on epithelial state and in the degree of corneal hypoesthesia.

Plasma rich in growth factors (PRGF-Endoret) represent a new technology using autologous proteins, growth factors and biomaterials as therapeutic formulations for different regenerative purposes. Under strict pharmaceutical development, it is possible to develop biologically stable eye drops, which have been shown to be useful for treating diverse ocular surface diseases. PRGF-Endoret eye drops could be an alternative therapy for patients with NK, and thus the objective of this clinical trial is to demonstrate its possible efficacy and its safety in patients with NK in stages 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over.
* With neurotrophic keratitis at stages 2 or 3 affecting only one eye.
* Persistent epithelial defect or corneal ulcer of at least 2 weeks duration resistant to one or more traditional non-surgical treatments .
* Corneal sensitivity reduction test in the area of the persistent epithelial defect or corneal ulcer and out of the defect area in at least one corneal quadrant.
* No objective clinical evidence of improvement in the two weeks prior to enrollment.
* Patients who have previously read and signed the informed consent.

Exclusion Criteria:

* Patients with neurotrophic keratitis stages 2 or 3 that affects both eyes.
* With active ocular infection or inflammation not related to the neurotrophic keratitis
* Any other eye disease that requires of topical ocular treatment in the affected eye during study.
* Patients with severe vision loss
* Patients with severe blepharitis and/or severe Meibomian glands disease
* History of eye surgery in the three months prior to enter the study, or patients who plan to undergo surgery.
* Having received previously surgical procedures for the treatment of NK.
* Use of therapeutic contact lenses or for refractive correction during study.
* Patients with punctual occlusion or insertion of punctual plugs previous to the study
* Evidence of corneal ulcer affecting the corneal stroma or cornea perforation.
* Presence of any disorder or ocular or systemic disease that could limit the treatment effectiveness or its evaluation,
* Any need of change (at that time or planned) in the dose of systemic drugs known to disrupt the functioning of the trigeminal nerve
* Known hypersensitivity to any of the procedural compounds (eg. fluoresceine).
* Presence of blood disorders associated with platelet disorders or clotting, or receiving anticoagulants drugs or antiplatelet agents.
* Patients with positive result in one of the serological tests for syphilis, Hepatitis B-C or AIDS I / II.
* Patient in current treatment for their pathology already well managed.
* Use of any investigational drug within 4 weeks prior to the screening visit.
* Pregnant women or intended to be pregnant.
* Participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-04 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a reduction of corneal defect of >50% | 4 weeks

SECONDARY OUTCOMES:
Percentage of patients with a reduction of corneal defect of >50% | 2 weeks
Percentage of patients showing complete healing of the corneal defect | 4 weeks
Percentage of patients showing complete healing of the corneal defect | 2 weeks
Measurement of the depth of the corneal defect (mm) | 2 and 4 weeks
Changes in percentage in Best corrected visual acuity (BCVA LogMAR) | 2 and 4 weeks
Ocular pain with VAS scale | 2 and 4 weeks
Osmolarity of lacrimal film | 2 and 4 weeks
Measurement of treatment tolerance | 2 and 4 weeks
  Measurement of treatment tolerance with a 0 4 score
Adverse events | 2 and 4 weeks
  Percentage of adverse event occurrence

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Instituto Clínico Quirúrgico de Oftalmología (ICQO), Bilbao, Bizkaia
  - Instituto Oftalmológico Fernández-Vega, Oviedo, Principality of Asturias
  - Instituto de Microcirugía Ocular (IMO), Barcelona
  - Hospital Ramón y Cajal, Madrid